CLINICAL TRIAL: NCT06453031
Title: Short-term Outcomes of Gastric Ischemic Preconditioning Before Esophagectomy With Preoperative Embolization of the Left Gastric Artery: A Prospective Single-Center Study
Brief Title: Gastric Ischemic Preconditioning Before Esophagectomy
Status: Active, not recruiting | Type: Observational
Sponsor: CHU Rennes - Hopital Pontchaillou (Other)
Responsible Party: Principal Investigator, LIVIN Marie, Chef de Clinique, CHU Rennes - Hopital Pontchaillou
Other Study IDs: CHU Pontchaillou Rennes
Record Dates: First submitted 2024-06-02; First posted 2024-06-11 (Actual); Last update posted 2024-06-11 (Actual); Status verified 2024-06

CONDITIONS: Operable Esophageal Cancer; Embolization of the Left Gastric Artery Prior to Surgery

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patient who underwent Gastric Ischemic Preconditioning Before Esophagectomy: Patient with operable esophageal cancer who underwent embolization of the left gastric artery prior to surgery
  Interventions: Procedure: Gastric Ischemic Preconditioning Before Esophagectomy

INTERVENTIONS:
Procedure: Gastric Ischemic Preconditioning Before Esophagectomy — Does embolization of the left gastric artery prior oesophagectomy reduce postoperative complications, particularly anastomotic leaks and ischemia of the gastric conduit?

SUMMARY:
The aim of the study is to investigate the impact of left gastric artery embolization before esophagectomy on postoperative complications, particularly anastomotic leaks and necrosis of the gastric conduit.

ELIGIBILITY:
Inclusion Criteria:

Patient with operable esophageal cancer who underwent embolization of the left gastric artery prior to surgery.

Exclusion Criteria:

Patient with no operable esophageal cancer

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patient with operable esophageal cancer who underwent embolization of the left gastric artery prior to surgery.
Sampling Method: Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2024-06-01 (Actual); Primary Completion 2025-06 (Estimated); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
Anastomotic leak | 6 months
Anastomotic stenosis | 6 months
Gastric conduit necrosis | 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- Livin, Rennes, Brittany Region, France